CLINICAL TRIAL: NCT03971552
Title: Gadolinium-Enhanced Extracranial MRA Prior to Mechanical Thrombectomy Is Not Associated With an Improved Procedure Speed
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 30687224
Record Dates: First submitted 2019-05-26; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Stroke
Keywords: Mechanical thrombectomy; Magnetic resonance angiography; Angiogram; Angiography; Magnetic resonance imaging; Revascularization
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: gadolinium-enhanced extracranial magnetic resonance angiogram — 288 of the 912 acute ischemic stroke patients received gadolinium-enhanced extracranial MRA additionally to the standardized stroke MRI imaging protocol.

SUMMARY:
The objective was to assess if performing a pre-intervention gadolinium-enhanced extracranial magnetic resonance angiogram (MRA) in addition to intracranial vascular imaging was associated with improved thrombectomy time metrics.

Consecutive patients (912) treated by mechanical thrombectomy (MT) at a large comprehensive stroke center between January 2012 and December 2017 who were screened using pre-intervention MRI were included. Patient's characteristics and procedural data were collected. Analyses were performed to compare mechanical thrombectomy speed, efficacy, complications, and clinical outcomes between patients with and without pre-intervention gadolinium-enhanced extracranial MRA.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke (AIS) patients who underwent magnetic resonance imaging (MRI) based screening for acute neurovascular evaluation and who underwent mechanical thrombectomy (MT) at one comprehensive stroke center.
Sampling Method: Non-Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
time from groin puncture to clot contact | 1 day
  in minute time from onset to recanalization complications [embolic or hemorrhagic]

SECONDARY OUTCOMES:
modified Rankin Score | 3 months

IPD SHARING:
Plan to Share IPD: No